CLINICAL TRIAL: NCT06824922
Title: Be Yourself" Educational Intervention With Web Page and Chatbot to Promote Self-determined Motivation and Prevent Teenage Pregnancy: Pilot Trial.
Brief Title: "Educational Intervention 'Be Yourself': Digital Innovation to Prevent Teenage Pregnancy"
Acronym: BYE-Chat
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Natanael Librado Gonzalez, Master of Science in Nursing, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Autonomous University of Nuevo; No. Registro: FAEN-D-2021 (Other: Autonomous University of Nuevo)
Record Dates: First submitted 2025-02-03; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Prevenir el Embarazo Adolescente
Keywords: Self-determination; Teenage Pregnancy; Sexual behaviour; Prevention; Randomized controlled trial
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Intervention Model Description: This Pilot Randomized Controlled Trial with a parallel intervention model, where one group receives the educational intervention "Be Yourself" and the other receives conventional sex education. It uses an Open Label design and has a preventive purpose (Prevention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Intervention "Be yourself" (Experimental): The experimental group will receive the educational intervention "Be Yourself", designed to prevent sexual risk in high school adolescents through self-determined motivation. This intervention is based on the MACSPEA model, competency-based learning and stages of change, and uses an interactive web page and a chatbot for follow-up and activities.
  Intervention: The intervention consists of three interactive educational sessions:
  Session One: Introduction to self-determined motivation and key aspects of sexuality, including anatomy, physiology, and sexual health.
  Session two: Exploration of sexual goals, values and communication, using role-plays and activities to strengthen decision-making and problem-solving skills.
  Third session: Focus on motivation for healthy decision making and prevention of pregnancy and STIs, with a follow-up session via website and chatbot.
  Duration: Each session lasts 60 minutes, for a total of 10 hours and 20 minutes of intervention.
  Interventions: Behavioral: "Be yourself", educational intervention with chatbot to promote self-determined motivation and prevent adolescent pregnancy: pilot trial protocol
- Control Group (CG) - Conventional Sex Education (Active Comparator): The control group will receive conventional sex education, which focuses on the transmission of knowledge about anatomy, physiology and contraceptive methods, as well as self-care of sexual health.
  Intervention: Two theoretical sessions of one hour each will be given:
  First session: orientation on sexual health, contraceptive methods and teen pregnancy prevention, through a PowerPoint presentation.
  Second session: Development of sexual health self-care skills, with emphasis on informed decision making and self-respect.
  Duration: Each session lasts 60 minutes, for a total of 2 hours of intervention.
  Interventions: Other: Conventional Sex Education

INTERVENTIONS:
Behavioral: "Be yourself", educational intervention with chatbot to promote self-determined motivation and prevent adolescent pregnancy: pilot trial protocol — The "Be Yourself" educational intervention stands out for its focus on self-determined motivation and teen pregnancy prevention. Unlike traditional interventions, which focus on transmitting information, this intervention promotes adolescent autonomy in making responsible sexual decisions. It uses interactive technology such as a web page and a chatbot, which provide personalized follow-up and reinforcement activities between sessions, encouraging active participation. It also employs competency-based learning, which strengthens practical and emotional skills, such as effective communication and problem solving. Sessions include role-plays and practical activities to apply what has been learned. This comprehensive approach and the use of digital platforms distinguish "Be Yourself" from other interventions, offering continuous and personalized accompaniment to reinforce learning throughout the process.
  Arms: Educational Intervention "Be yourself"
Other: Conventional Sex Education — For the CG, two theoretical sessions are planned. In the first, an orientation on adolescent sexual health will be provided through a one-hour PowerPoint presentation. Topics of anatomy, physiology, biological changes in adolescence and contraceptive methods will be addressed, highlighting their proper use and the prevention of adolescent pregnancy. The second session, also lasting one hour, will develop sexual health self-care skills, discussing the importance of self-care, self-respect and informed decision making. There will be a question and answer session to address concerns and reflect on how self-care contributes to a healthy and safe sexual life.
  Arms: Control Group (CG) - Conventional Sex Education

SUMMARY:
Introduction: Adolescent pregnancy and early initiation of sexual activity is a serious global public health problem, every year, around sixteen million adolescents between 15 and 19 years of age give birth, representing 11% of all births globally. Objective: To design a protocol of a pilot Randomized Controlled Trial to evaluate the preliminary efficacy of the "Be Yourself" intervention to increase self-determined motivation to prevent pregnancy in adolescents in secondary education. Methods: The protocol was developed based on the Protocol Items: ecommendations for Interventional Trials 2013 (SPIRIT2013) Statement, in the City of Monterrey, Nuevo León, Mexico in 2023. Results: The protocol outlined the design of the intervention, structured the content of the sessions using a logic model of intervention, and developed manuals for program facilitators and guides for participants. In addition, a website and a chatbot with Artificial Intelligence were developed, and the strategy for the application of the evaluation instruments was established. Conclusion: The educational intervention "Be yourself" is projected as a promising program to promote self-determined motivation and prevent adolescent pregnancy.

DETAILED DESCRIPTION:
Background and Rationale Adolescent pregnancy is a critical global public health issue, with approximately 16 million adolescents aged 15 to 19 giving birth each year, accounting for 11% of all global births. This phenomenon significantly impacts maternal and child health, as well as the social and economic well-being of young mothers and their families. In Mexico, adolescent pregnancy rates remain among the highest globally, with more than 90% of new sexually transmitted infections (STIs) occurring in young women, and significant disparities in fertility rates between rural (2.8) and urban (2.01) areas.

Several studies have identified key risk factors associated with adolescent pregnancy, including lack of knowledge about contraception, low risk perception, peer pressure, low self-esteem, and limited communication about sexuality. Additionally, many traditional interventions have been limited in scope and effectiveness, as they fail to integrate motivational approaches or technological tools that align with adolescent communication preferences.

To address these challenges, the "Be Yourself" educational intervention was designed based on Self-Determination Theory and behavioral change models, aiming to foster self-determined motivation for adolescent pregnancy prevention. The intervention incorporates innovative strategies, including an artificial intelligence-powered chatbot and a web-based platform, allowing for dynamic, interactive, and accessible learning experiences for adolescents.

General Objective:

To evaluate the preliminary efficacy of the "Be Yourself" intervention in increasing self-determined motivation and promoting preventive behaviors against adolescent pregnancy among secondary school students.

Specific Objectives:

1. Assess the intervention's impact on adolescents' self-determined motivation.
2. Evaluate changes in knowledge regarding sexual and reproductive health.
3. Measure improvements in communication about sexuality with parents, friends, and partners.
4. Determine the acceptability and feasibility of using a chatbot for sexual health education.
5. Examine changes in behavioral intentions and pregnancy prevention behaviors. Study Design This study follows a pilot randomized controlled trial (RCT) with a pretest-posttest design, comparing the "Be Yourself" educational intervention to a traditional sexual education program.

Participants and Inclusion Criteria:

* Adolescents aged 12 to 15 enrolled in public secondary schools in Santa Catarina, Nuevo León, Mexico.
* Access to the internet to participate in the web-based platform.
* Parental consent and adolescent assent obtained.
* No prior participation in similar programs in the last six months.

Exclusion Criteria:

* Adolescents are diagnosed with psychological or cognitive disorders that interfere with comprehension.
* Current pregnancy.

Sample Size and Sampling Procedure:

The study will recruit 150 participants, randomly assigned in a 1:1 ratio to the following groups:

* Experimental Group (EG): Receives the "Be Yourself" intervention, including interactive sessions, chatbot support, and access to the web platform.
* Control Group (CG): Receives conventional sexual education through lecture-based sessions.

Participants will be randomly selected, accounting for a 20% dropout rate. Description of the "Be Yourself" Intervention The intervention consists of three interactive educational sessions, combining theoretical and practical strategies in an innovative digital environment.

Intervention Components:

1. AI-Powered Chatbot: Answers sexual health questions, provides reminders, and encourages participation.
2. Web-Based Platform: Offers multimedia resources, interactive activities, and discussion forums.
3. Educational Sessions: Based on the Self-Determination Model for Adolescent Pregnancy Prevention.

Session Structure:

* Session 1: Introduction to self-determined motivation and self-awareness.
* Session 2: Strategies for responsible decision-making and assertive communication.
* Session 3: Goal setting and pregnancy prevention planning. Variables and Measurements

Validated instruments with high reliability coefficients (Cronbach's alpha ranging from 0.77 to 0.95) will be used to evaluate:

1. Primary Variables:

   * Self-determined motivation for pregnancy prevention.
   * Change in sexual and reproductive health knowledge.
2. Secondary Variables:

   * Communication about sexuality with parents, friends, and partners.
   * Behavioral intention for pregnancy prevention.
   * Level of satisfaction and engagement with the intervention. Assessments will be conducted at three time points: pretest, posttest, and a 3-month follow-up.

Data Analysis

The SPSS v26.0 software will be used for statistical analysis:

1. Descriptive Analysis: Means, standard deviations, and frequencies.
2. Normality Test: Kolmogorov-Smirnov test to determine data distribution.
3. Pretest-Posttest Comparisons:

   * Paired t-test (parametric variables).
   * Mann-Whitney U test (non-parametric variables).
4. Repeated Measures ANOVA to analyze changes over time. A significance level of p < 0.05 will be considered. Ethical Considerations

   * The study has been approved by the Ethics Committee of the School of Nursing at the Universidad Autónoma de Nuevo León.
   * Parental consent and adolescent assent will be obtained.
   * Confidentiality will be ensured through anonymous participant ID codes.
   * Participation is voluntary, with the option to withdraw at any time without consequences.

Expected Outcomes

The "Be Yourself" intervention is expected to:

1. Increase adolescents' self-determined motivation.
2. Enhance knowledge of sexual health and pregnancy prevention.
3. Improve communication about sexuality with parents and peers.
4. Strengthen behavioral intentions regarding contraception and pregnancy planning.
5. Increase acceptance of digital strategies for health education.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 11 and 15 years of age enrolled in public high schools in Nuevo León will be included.

public high schools in Nuevo León.

* Be male or female, regardless of whether they have initiated their sexual life. sexually active.
* Have access to a computer room with internet to use the web page and the interventions chatbot.

the interventions chatbot.

* Live at the same address with their parents or legal guardian.

Exclusion Criteria:

* Have previously participated in a similar sexuality intervention.
* Have cognitive or developmental difficulties that impede their understanding of the intervention and use of the technology platform, including people with
* Autism Spectrum Disorder (ASD) at levels that affect functional communication, Attention Deficit Hyperactivity Disorder (ADHD) with severe attention difficulties, or those who cannot read and write.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-02-06 (Estimated); Primary Completion 2025-04-06 (Estimated); Study Completion 2025-06-06 (Estimated)

PRIMARY OUTCOMES:
Increased rates of Self-Determined Motivation to prevent teenage pregnancy | It will be evaluated before the intervention (pretest 1), after completing the intervention (posttest 2) and 3 months after follow-up.
  Change in levels of self-determined motivation for adolescent pregnancy prevention will be assessed using context-specific psychometric tools. It is expected that the intervention will increase intrinsic motivation and encourage responsible sexual decision-making.
  For this measurement, the Behavioral Regulation in Exercise Questionnaire (BREQ-3), originally developed to assess motivation in physical activity and subsequently adapted to the Mexican context to measure behavioral regulation in pregnancy prevention, will be used. The peer-reviewed adaptation retained its psychometric validity.
  The questionnaire uses a five-point Likert scale and calculates self-determined motivation using the Self-Determination Index (SDI) with the following formula: 3 * intrinsic regulation) + (2 * integrated regulation) + (1 * identified regulation) - (1 * introjected regulation) - (2 * external regulation) - (3 * no motivation), with reliability reported in different studies.
Increase in the Level of Knowledge about Pregnancy Prevention | It will be evaluated before the intervention (pretest 1), after completing the intervention (posttest 2) and 3 months after follow-up.
  The Sexual and Reproductive Health Knowledge Scale will be used to assess the level of knowledge in this area. The instrument, originally composed of 128 items, addresses four dimensions: sexual health, reproductive health, HIV/AIDS and STIs, and condom use. For this study, 29 items were selected from the dimensions of sexual health, reproductive health and condom use.
  The responses follow a Likert-type scale with options: true (1), false (2) and don't know (8), although in some items the "true" and "false" scores are reversed. For the analysis, the "don't know" option will be recoded as 0, and the correct answers as 1, establishing a dichotomous scale (0-1), where higher scores indicate a higher level of knowledge.
Improving Communication on Sexual Issues | It will be evaluated before the intervention (pretest 1), after completing the intervention (posttest 2) and 3 months after follow-up.
  This outcome will be assessed using the Communication about Sexual Issues with Parents, Friends, and Partners Instrument, focusing on pregnancy prevention. Six of the original nine items will be used. The response scale is a five-point Likert scale (1 = not at all, 5 = very much), with a total score from 6 to 30, where higher values indicate greater perceived communication.
  The information received on reproduction, contraception, condom use and social pressure in sexual relations will be analyzed. An increase in the quality and frequency of these interactions is expected, favoring informed decision making.
Change in Life Goals | It will be evaluated before the intervention (pretest 1), after completing the intervention (posttest 2) and 3 months after follow-up.
  The Aspirations Index Instrument will be used to evaluate the importance of life goals in adolescents, considering both extrinsic goals (wealth, fame, image and power) and intrinsic goals (relationships, personal growth, social contribution, self-expression and mastery).
  The questionnaire, previously adapted to the Mexican context, will have 51 items and will be applied using a seven-point Likert scale (1 = not at all important, 7 = very important). Higher scores will reflect a greater importance given to personal aspirations.
  It is expected that the application of this instrument will provide reliable results, supported by previous studies that have reported.
Satisfaction of Basic Psychological Needs: autonomy, relationships and competence. | It will be evaluated before the intervention (pretest 1), after completing the intervention (posttest 2) and 3 months after follow-up.
  The Basic Psychological Needs Satisfaction and Frustration Scale (BPNSFS) will measure adolescents' perceptions of satisfaction and frustration of their needs for autonomy, competence and relationships in the context of pregnancy prevention.
  The instrument uses a Likert scale from 1 (totally false) to 5 (totally true), where higher satisfaction scores indicate greater well-being, while higher frustration scores reflect greater discomfort.
  For this study, the version adapted and validated in adolescents will be used, with high correlations in satisfaction and frustration, which supports its internal consistency and validity in the measurement of these factors.

SECONDARY OUTCOMES:
Risk and Protective Intention | It will be evaluated before the intervention (pretest 1), after completing the intervention (posttest 2) and 3 months after follow-up.
  The Adolescent Sexual Activity Intention Scale will assess the willingness of both female and male adolescents to adopt protective or risky behaviors in their sexual lives. This measure is derived from the Female and Male Reproductive Sexuality Questionnaires (F-M CSR), developed to identify factors such as personal attitudes, normative beliefs, and perceived control in sexual decision making.
  The scale consists of six items, organized into two categories: risk intention and intention towards protection, addressing the use of contraceptive methods, abstinence and delaying the onset of sexual activity. A Likert scale from 1 (strongly disagree) to 5 (strongly agree) is used, where higher values indicate a greater intention to adopt the evaluated behavior.
  Examples of items include: "When I have sex, I plan to use condoms to prevent pregnancy and STIs" (male version) and "When I have sex, I plan to take oral pills to prevent pregnancy" (female version).
Sexual behavior in relation to teenage pregnancy prevention. | It will be evaluated before the intervention (pretest 1), after completing the intervention (posttest 2) and 3 months after follow-up.
  The sexual behavior variable in relation to the prevention of adolescent pregnancy will be measured using the Sexual Activity Scale, adapted to evaluate this behavior in the context of adolescent pregnancy prevention. This scale measures the frequency of five behaviors: holding hands, kissing, touching, caressing genitals and having sexual intercourse, using a Likert scale from 1 (never) to 5 (always).
  From this assessment, three indicators will be generated: conventional, pre-penetrative and penetrative sexual activity. In addition, risk factors such as age of sexual debut, number of partners, frequency of penetrative sex, condom use and perceived risk of pregnancy will be analyzed.
  For sexually inexperienced adolescents, their willingness to initiate sexual intercourse will be explored by means of statements evaluated on a scale of 1 to 5, where higher scores will indicate a greater inclination towards sexual activity.
Pregnancy prevention sexual behavior Pregnancy | It will be evaluated before the intervention (pretest 1), after completing the intervention (posttest 2) and 3 months after follow-up.
  The scale used to measure pregnancy-preventive sexual behavior is based on the Sexual Health and Reproductive Health Knowledge Scale, derived from Vargas' (2013) Psychometric Scale of Knowledge, Attitudes and Practices in Sexual Health and Reproductive Health. This scale includes four dimensions: sexual health, reproductive health, HIV/AIDS and STIs, and condom use, each subdivided into knowledge, attitudes, and practices. For this study, 20 items were selected from the dimensions of sexual health, reproductive health, and condom use, focusing on the category of practices.
  The scale uses a Likert-type response with five options: always = 1, almost always = 2, sometimes = 3, almost never = 4, and never = 5. However, items 1, 5, 10, 12 and 19 have inverted scores. The lower the score, the greater the manifestation of pregnancy prevention behavior.
Process of sexual behavior change in adolescents | It will be evaluated before the intervention (pretest 1), after completing the intervention (posttest 2) and 3 months after follow-up.
  The University of Rhode Island Change Assessment Scale (URICA) will be adapted to measure the Adolescent Sexual Behavior Change Process. This adaptation will assess the phases of change - precontemplation, contemplation, action, and maintenance - as they relate to adolescent sexual behavior, using a 5-point Likert scale. The items of the instrument will be adjusted to be relevant and specific to the context of adolescent sexuality, thus allowing for an accurate assessment of readiness to change in this population. The score obtained will be calculated by averaging the items in each phase, and the formula for determining readiness to change in relation to sexual behavior will be used.
  The formula for calculating readiness to change on the University of Rhode Island Change Assessment Scale (URICA) is as follows:
  Readiness to Change = (Mean Contemplation + Mean Action + Mean Maintenance) - Mean Precontemplation.

OTHER OUTCOMES:
Evaluation of System Usability in the "Be Yourself" Intervention | Perceived usability of the 'Be Yourself' website and its chatbot will be assessed at the end of the intervention group sessions (around week 8), and again at the 3-month follow-up (approximately week 20).
  The System Usability Scale (USS) will be used to evaluate the perceived usability of the web platform and chatbot of the "Be Yourself" intervention. This scale consists of 10 items, with both positive and negative statements, and its total score ranges from 0 to 100, where higher values indicate better usability. The EUS measures two main factors: "Usability" (items 1, 2, 3, 5, 6, 7, 8 and 9) and "Ease of Learning" (items 4 and 10).
  In this evaluation, aspects such as ease of use, integration of functions, consistency in navigation and user confidence when interacting with the platform and the chatbot will be analyzed. The results will allow us to identify areas for improvement, optimize the participants' experience and strengthen the accessibility of the educational intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Natanael Librado González, Master, Principal Investigator — Universidad Autónoma de Nuevo León
Locations (1):
- Autonomous University of Nuevo Leon, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to strict ethical and confidentiality considerations. The study complies with current personal data protection regulations, guaranteeing the privacy and security of the information of the adolescent participants. The results will be presented only in aggregated and anonymized form, avoiding any possibility of identification. In addition, the informed consent signed by the participants and their legal guardians does not contemplate the disclosure of individual data to third parties.

REFERENCES:
- [Background] Ryan RM, Deci EL. Self-Determination Theory: Basic Psychological Needs in Motivation, Development, and Wellness. Guilford Publications; 2018.
- Available data/document: Study Protocol: Protocolo_ECA_piloto — https://drive.google.com/file/d/1PhNe1G9PVs2FkOmKeyXazMLW3l-sxRR7/view?usp=sharing

DOCUMENTS (1):
  • Study Protocol (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT06824922/Prot_000.pdf